CLINICAL TRIAL: NCT06950372
Title: Rebound Pain After Volar Plate Surgery in Infraclavicular Brachial Plexus Block With Ropivacaine 3.75 mg/ml Compared With 7.5 mg/ml. A Prospective, Parallelgroup, 2-arm, Triple Blinded Randomised Controlled Trial
Brief Title: Ropivacaine Concentration and Rebound Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Anette Aasen, Principal Investigator, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU CT 2024-514795-41-00; 2024-514795-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-26; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Radius Fracture Distal; Rebound Pain
Keywords: Rebound pain; Peripheral nerve block; Distal radius fracture; Brachial plexus block; Ropivacaine
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low concentration (Experimental): Ropivacaine 3.75 mg/ml
  Interventions: Drug: Ropivacaine concentration low
- High concentration (Active Comparator): Ropivacaine 7.5 mg/ml
  Interventions: Drug: Ropivacaine concentration high

INTERVENTIONS:
Drug: Ropivacaine concentration low — Brachial plexus nerve block with ropivacaine 3.75 mg/ml
  Arms: Low concentration
Drug: Ropivacaine concentration high — Brachial plexus nerve block with ropivacaine 7.5 mg/ml
  Arms: High concentration

SUMMARY:
The goal of this clinical trial is to see if the concentration of a local anesthetic (ropivacaine) in peripheral nerve block is related to the severness of pain after surgery of distal radius fractures in adults.

The main questions it aims to answer are:

* Is concentration of ropivacaine related to severeness, duration and type of postoperative pain?
* Is concentration of ropivacaine related to analgetic consumption after surgery?
* Is concentration of ropivacaine related to block sucess rate during surgery and patient satisfaction after surgery?

Researchers will compare ropivacaine 3.75 mg/ml and 7.5 mg/ml used in brachial plexus peripheral nerve block. Participipants are randomized to one of the two concentrations. The peripheral nerve block is standard anesthetic treatment for distal radius fractures scheduled for volar plate surgery at Oslo University Hospital. All other treatment for the condition will be the same as standard treatment.

Participants will answer a questionnaire regarding pain, physical function, medication and life quality at different points of time after surgery, up to 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal radius fracture, scheduled for volar plate surgery
* Surgery up to 20 days after fracture trauma
* 18 to 80 years old (inclusive)
* ASA 1, 2 or stable ASA 3
* Body Mass Index (BMI) 18 to 40 kg/m2 (inclusive)
* Weight of 50 kg or more
* Ability to communicate sufficiently in a scandinavian language
* Capable of giving a signed informed consent
* Ability and willingness to understand og be compliant to the study

Exclusion Criteria:

* Contemporaneous painful injuries
* Existing long-term pain
* Peripheral nerve damage in the arm with radius fracture
* Patients who prior to fracture trauma use opioids, psycothropic drugs or medication, with or without prescription, with significantly sedative effect on regular basis.
* Excessive use of alcohol (more than 15 units of alchol per week for men, more than 8 units of alchol per week for women, or patients reporting to be incapable of avoiding alcohol as long as they use strong opioids).
* Progressive neurologic disease (inclusive diabetic neuropathy).
* Skin infection at the site for brachial plexus nerve block
* Other contraindications for brachial plexus nerve block
* Contraindications for ropivacaine, paracetamol, etoricoxib, dexamehtasone or oxycodone
* Previous allergic reaction to local anaesthetics or etoricoxib, dexamethasone, oxycodone or paracetamol.
* Pregnant or breast-feeding women at surgery day (they do not get excluded if they become pregnant in the follow up period after intervention and surgery)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Worst pain score during the first 48 hours after surgery | 48 hours after end of surgery
  Pain score on Verbal Numeric Rating Scale (VNRS) from 0 to 10, where 0 represents no pain at all and 10 represents worst pain imaginable.

SECONDARY OUTCOMES:
Rebound pain | From end of surgery until nerve block resolution, normally within the first 48 hours after surgery.
  Number of patients reporting pain score on Verbal Numeric Rating Score (VNRS) of 7 or higher at nerve block resolution, where 0 represents no pain at all and 10 represents worst pain imaginable.
Pain score at different points of time after surgery | From baseline, end of surgery, until 6 weeks after surgery.
  Pain score 0 to 10 on Verbal Numeric Rating Score (VNRS), where 0 represents no pain at all and 10 represents worst pain imaginable. Pain Score (VNRS 0-10) measured in the Post Anaesthesia Care Unit (PACU) and at 4 hours, 8 hours, 24 hours, 48 hours, 3 days, 7 days and 6 weeks after surgery.
Duration of moderate and strong pain | From baseline, end of surgery, until first time patient reports VNRS below 7 and/or 4, normally within the first 48 hours.
  Pain measured on Verbal Numeric Rating Score (VNRS) from 0 to 10, where 0 represents no pain at all and 10 represents worst pain imaginable.
  Duration of moderate pain, defined as time from VNRS above or equal to 4, after block resolution to first time patient reports VNRS below 4.
  Duration of strong pain, defined as time from VNRS above or equal to 7, after block resolution to first time patient reports VNRS below 7.
Average and worst pain experience after surgery at different points of time | From baseline, end of surgery, until 7 days after surgery.
  Pain measured on Verbal Numeric Rating Score (VNRS) from 0 to 10, where 0 represents no pain at all and 10 represents worst pain imaginable.
  Average pain score (VNRS 0-10) at 8-24 hours after surgery, 24-48 hours after surgery, last 24 hours at 3 days and 7 days after surgery.
  Worst pain score (VNRS 0-10) at 8-24 hours after surgery, 24-48 hours after surgery, last 24 hours at 3 days and 7 days after surgery.
Long-lasting pain | From baseline, end of surgery, until 6 weeks after surgery.
  Pain measured on Verbal Numeric Rating Score (VNRS) from 0 to 10, where 0 represents no pain at all and 10 represents worst pain imaginable.
  Pain score (VNRS 0-10) at rest and with movement of arm at 6 weeks after surgery.
  Worst pain (VNRS 0-10) during last week at 6 weeks after surgery.
  Average pain (VNRS 0-10) during last week at 6 weeks after surgery.
Analgesic consumption after surgery | From baseline, end of surgery, until 6 weeks after surgery.
  Total opioid consumption, measured in oral morphine equivalent, first 8 hours, first 24 hours, 24-48 hours, 48-72 hours, 72 hours to 1 week and last week at 6 weeks after surgery.
  Total analgesic consumption at the same times as above.
Duration of motoric and sensoric nerve block | From intervention, peripheral nerve block (needle out), until motoric and sensory resolution of nerve block, normally within the first 48 hours after intervention.
  Duration of motoric block: Time from nerve block (needle out) to first time the patient can hold an item with the blocked arm and lift i to the mouth area.
  Duration of sensory block: Time from nerve block (needle out) to first sensation of pain.
  We will also register time from nerve block (needle out) to first rescue analgesic.
Life quality | From baseline, end of surgery, until 6 weeks after surgery
  Estimation of pain burden with different quality of life measures at different time points after surgery:
  Quality of sleep, work ability, social life and cognitive function using Likert Scale.
  Number of patients answering "yes" to the question: "Do you have bothersome pain?".
  Measures registered 24 hours, 48 hours, 72 hours, 1 week and 6 weeks after surgery.
Quality of long-term pain | 6 weeks after baseline, intervention and surgery.
  If long-term pain, what type of pain is experienced (heat, cold, burning, prickly, tingling, itchy, squeezing). Registration of pain quality without direct stimulation and after direct stimulation in surgery area and 5-10 cm away from surgery area.
Patient satisfaction | From enrollment until 6 weeks after surgery
  Yes or no to the question; "Are you satisfied with the pain treatment?"
Block success rate | From intervention, when nerve block is performed, until 2 hours after surgery.
  Try to estimate if there is a difference in block success rate between the two concentrations. Sensory and/or motor test of relevant nerves (musculocutaneous, radial, median, ulnar and medial antebrachial cutaneus nerve) before surgery (45 minutes after nerve block and repeated if necessary) and in Post Anesthesia Care Unit (PACU) after surgery.
  In addition, yes or no to the question; "Was the block adequate for surgery?" (Registered by anaesthetic personell during surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Anette Aasen, MD, Anesthesiologist, Principal Investigator — University of Oslo and Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after deidentification, will be available in Norwegian at a request. In addition, the Study Protocol is a public document from application moment. Researchers who provide a methodologically sound proposal will receive access to the deidentified individual pariticipant data, to achieve aims in the approved proposal. The data will be available immediately following publication and ending 5 years following article publication. Proposals should be directed to anette.aasen@medicin.uio.no.